CLINICAL TRIAL: NCT07129863
Title: Caffeine Mouth Rinsing at Different Doses Does Not Enhance Anaerobic Sprint Performance in Female Team-Sport Athletes: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Caffeine Mouth Rinsing at Different Doses in Female Team-Sport Athletes: A Randomized, Double-Blind, Placebo-Controlled Trial
Acronym: MORISINGFEMALE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia Comillas (Other)
Collaborators: Eastern Mediterranean University (Other); Northumbria University (Other); Universidad Francisco de Vitoria (Other); Ankara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UPC-Comillas
Record Dates: First submitted 2025-08-11; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Dietary Supplement; Sports Performance
Keywords: carbohydrate; nutrition; mouth rinse; placebo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (water) (Placebo Comparator): Placebo: Mouth rinse with plain water, containing no caffeine, serving as the control condition.
  Interventions: Dietary Supplement: Placebo: Mouth rinse with plain water
- Low mouth rinse caffeine concentration (Experimental): Low caffeine concentration: Mouth rinse containing 1% caffeine solution (based on weight/volume).
  Interventions: Dietary Supplement: Experimental: Low mouth rinse caffeine concentration (1%)
- Moderate mouth rinse caffeine concentration (Experimental): Moderate caffeine concentration: Mouth rinse containing 2% caffeine solution (based on weight/volume).
  Interventions: Dietary Supplement: Moderate caffeine concentration (2% caffeine solution weight/volume).
- High mouth rinse caffeine concentration (Experimental): Moderate caffeine concentration: Mouth rinse containing 3% caffeine solution (based on weight/volume).
  Interventions: Dietary Supplement: High caffeine concentration (3% caffeine solution weight/volume).

INTERVENTIONS:
Dietary Supplement: Placebo: Mouth rinse with plain water — Placebo: Mouth rinse with plain water, containing no caffeine, serving as the control condition.
  Arms: Placebo (water)
Dietary Supplement: Experimental: Low mouth rinse caffeine concentration (1%) — Arm Description: Low caffeine concentration: Mouth rinse containing 1% caffeine solution (based on weight/volume).
  Arms: Low mouth rinse caffeine concentration
Dietary Supplement: Moderate caffeine concentration (2% caffeine solution weight/volume). — Moderate caffeine concentration: Mouth rinse containing 2% caffeine solution (weight/volume).
  Arms: Moderate mouth rinse caffeine concentration
Dietary Supplement: High caffeine concentration (3% caffeine solution weight/volume). — High caffeine concentration: Mouth rinse containing 3% caffeine solution (weight/volume).
  Arms: High mouth rinse caffeine concentration

SUMMARY:
Objective:

To evaluate the effects of different caffeine mouth rinse concentrations (1%, 2%, and 3%) on Running Anaerobic Sprint Test (RAST) performance in female team-sport athletes.

Main Questions:

1. Do caffeine mouth rinses improve RAST performance in female team-sport athletes?
2. Do different caffeine mouth rinse concentrations affect ratings of perceived exertion (RPE)?

Method:

Thirteen trained female football and handball players (23.0 ± 4.5 years) completed four randomized, double-blind, crossover conditions (1%, 2%, and 3% caffeine mouth rinses, and placebo). Each trial involved six 35 m sprints separated by 10 s of rest. RPE was recorded immediately after each session.

DETAILED DESCRIPTION:
Objective:

To evaluate the acute effects of different caffeine mouth rinse concentrations (1%, 2%, and 3%) on anaerobic sprint performance and perceived exertion in trained female team-sport athletes. The study sought to determine whether this non-ingestive ergogenic strategy could enhance high-intensity running performance and reduce effort perception.

Main Questions:

1. Do different caffeine mouth rinse concentrations improve Running Anaerobic Sprint Test (RAST) performance in trained female team-sport athletes?
2. Do caffeine mouth rinses at varying concentrations influence ratings of perceived exertion (RPE) compared with placebo?

Is there an optimal caffeine concentration that balances potential performance benefits with reduced perceived exertion?

Method:

Thirteen trained female athletes (mean age 23.0 ± 4.5 years) competing in football and handball participated in a randomized, double-blind, placebo-controlled, crossover trial. Each athlete completed four experimental conditions: placebo, 1% caffeine mouth rinse, 2% caffeine mouth rinse, and 3% caffeine mouth rinse. In each session, participants performed a Running Anaerobic Sprint Test (RAST) consisting of six maximal 35 m sprints separated by 10 seconds of passive recovery. The RPE was assessed immediately after each test using a 1-10 scale.

ELIGIBILITY:
Inclusion Criteria

* Female team sports athletes aged between 18 and 35 years.
* Currently engaged in team sports.
* Non-smoker.

Exclusion Criteria

* Participants were excluded if they met any of the following conditions.
* Presence of a musculoskeletal injury within the six months prior to the study.
* Current smoker.
* Use of nutritional supplements or ergogenic aids that could influence sprint running performance (e.g., beta-alanine, creatine).
* Use of oral contraceptives.
* Known allergy to caffeine.
* Failure to meet the training requirement of at least six hours of team-based practice, a minimum of three days per week, over the past year.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2023-09-24 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Running-based anaerobic sprint test (RAST protocol) | 2-week
  The RAST was comprised of six 35 m sprints at maximum effort, each of which was followed by a 10 s passive rest period (including deceleration phase). Participants rinsed the solution in the final 5 s of the rest period accompanied by the counting of the tester, and then sprint back to the first timing gate with "GO" command. This was repeated until six sprints had been accomplished. Participants began to sprint running for a maximum of one step before the timing gate and were instructed not to decelerate before passing through the timing gate. Using a system of photocells (Newtest Powertimer 300-series, Newtest Oy, Tyrnävä, Finland), which was placed at the beginning and the end of the 35 m, the duration of each 35 m sprint running time was recorded. Using time of each sprint attempt, 1-) fastest sprint time, 2-) mean sprint time, and 3-) fatigue index were recorded

SECONDARY OUTCOMES:
Rating of perceived exertion (RPE) | 2-weeks
  Perceived exertion during each trial was assessed immediately after the Running Anaerobic Sprint Test (RAST) using a 1-10 numerical scale points, where:
  1 = Very, very light effort (minimal exertion, easy to continue)
  2-3 = Light effort (comfortable, mild strain)
  4-5 = Moderate effort (noticeable breathing and muscle activation)
  6-7 = Hard effort (challenging but sustainable for a short time)
  8-9 = Very hard effort (significant discomfort, near maximal effort)
  10 = Maximal effort (unable to continue beyond current level, exhaustion)
  This scale provided a subjective measure of the athletes' internal load, complementing the objective performance metrics from the sprint test.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Mersin, SBF C 116, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will be shared if previously is required